CLINICAL TRIAL: NCT00546741
Title: Pharmacokinetic Drug Interaction Study With Dapagliflozin and Metformin in Healthy Subjects
Brief Title: Drug Interaction With Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MB102-026
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Healthy Male and Female Subjects
Keywords: Diabetes,NOS
MeSH Terms: conditions — Diabetes Mellitus | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Dapagliflozin
- 2 (Active Comparator)
  Interventions: Drug: Metformin
- 3 (Active Comparator)
  Interventions: Drug: Dapagliflozin + Metformin

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 20 mg, once daily single dose
  Arms: 1
Drug: Metformin — Tablets, Oral, 1000 mg, once daily, single dose
  Arms: 2
Drug: Dapagliflozin + Metformin — Tablets, Oral, once daily, single dose
  Dapagliflozin: 20 mg
  Metformin: 1000 mg
  Arms: 3

SUMMARY:
The purpose of the study is to determine the effect of metformin on dapagliflozin exposure and the effect of dapagliflozin on metformin exposure in healthy volunteers. Additionally, the safety and tolerability of dapagliflozin will be assessed in the presence and absence of metformin in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, ages 18-45 with a body mass index of 18-32 kg/m2

Exclusion Criteria:

* Unwilling to use acceptable method of birth control
* current or recent (within 1 month) smoker
* abnormal liver function tests
* presence of edema
* history of diabetes mellitus
* history of heart failure or renal insufficiency
* history of chronic or recurrent urinary tract infections, or vulvovaginal mycotic infections
* history of Hepatitis C

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To determine the effect of metformin on the exposure of dapagliflozin and the effect of dapagliflozin on the exposure of metformin in healthy subjects after a single dose of each treatment | measures taken daily throughout the study

SECONDARY OUTCOMES:
To assess the safety and tolerability of dapagliflozin when administered alone or with metformin after a single dose of each treatment | measures will be taken at the beginning and end of the study, as well as 1 time every 3 days (Day -1 of each study period)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol-Myers Squibb Clinical Pharmacology Unit, Hamilton, New Jersey, United States

REFERENCES:
- See also: MB102026 _Redacted _CSR _synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3638&filename=MB102026%20_Redacted%20_CSR%20_synopsis.pdf